CLINICAL TRIAL: NCT06398652
Title: Comparative Study of the Efficacy, Safety, and Immunogenicity of CMAB015 and Secukinumab in Adult Patients With Moderate-severe Chronic Plaque Psoriasis
Brief Title: Comparative Study of CMAB015 and Secukinumab for Patients With Moderate to Severe Plaque Psoriasis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Taizhou Mabtech Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMAB015-002
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): CMAB015
  Interventions: Biological: CMAB015
- Active Comparator Arm (Active Comparator): Secukinumab
  Interventions: Biological: Secukinumab

INTERVENTIONS:
Biological: CMAB015 — Patients would receive 300 mg CMAB007 subcutaneous injections at week 0, 1, 2, 3, 4, 8 as induction therapy. Patients who obtain a 75% improvement relative to baseline in PASI scores would receive 300 mg CMAB007 subcutaneous injections every 4 weeks as maintain therapy, until the last treatment at week 48.
  Arms: Experimental Arm
Biological: Secukinumab — Patients would receive 300 mg secukinumab subcutaneous injections at week 0, 1, 2, 3, 4, 8 as induction therapy. Patients who obtain a 75% improvement relative to baseline in PASI scores would receive 300 mg secukinumab subcutaneous injections every 4 weeks as maintain therapy, until the last treatment at week 48.
  Other Names: Cosentyx
  Arms: Active Comparator Arm

SUMMARY:
The goal of this trial is to assess whether the efficacy of CMAB015 is similar to that of Secukinumab in patients with moderate-severe chronic plaque psoriasis. It will also learn about the similarity of CMAB015 and Secukinumab in terms of safety and immunogenicity in patients with moderate-severe chronic plaque psoriasis. The main question it aims to answer is:

In subjects with moderate to severe plate psoriasis treated with CMAB015, Is the proportion of patients achieving a 75% improvement in PASI (Psoriasis area and severity index) scores relative to baseline (PASI 75) the same as those treated with Secukinumab?

Participants will:

Receive treatment with 300 mg CMAB015 or Secukinumab by subcutaneous injection at weeks 0, 1, 2, 3, 4, and 8, followed by every 4 weeks until week 48.

Visit the clinic at weeks 0, 1, 2, 3, 4, and 8, followed by every 4 weeks until week 52.

Be evaluated with PASI scores, body surface area (BSA) scores and investigator's global assessment (IGA) (mod 2011) scores.

DETAILED DESCRIPTION:
This study was a multicenter, randomized, double-blind, secukinumab controlled, 1:1 ratio parallel grouping, equivalent design. The study treatment period would be 52 weeks, including a 12-week induction therapy period and a 40-week maintenance therapy period. The primary endpoint was the proportion of patients achieving at least a 75% improvement in PASI scores from baseline at 12 weeks, with an equivalence cut-off of ±15%. A total of 336 adult patients with moderate-to-severe plaque psoriasis are planned to be enrolled, with 168 cases in each group. Eligible subjects received 300 mg CMAB015 or Secukinumab subcutaneous injection. Patients who do not achieve at least a 50% improvement in PASI scores at week 12 would withdraw from the study, and patients who achieve a 50% improvement continue on maintenance therapy until the last treatment at week 48.

This study is a double-blind design, and a central randomization system woud be used to randomize subjects. The control factors for randomization are body weight (<60 kg, ≥60 kg), prior treatment (prior systemic therapy with no prior biologics, prior systemic therapy with biologics), concomitant psoriatic arthritis (yes, no), and PK intensive sampling (yes, no).

ELIGIBILITY:
Inclusion Criteria:

* History of confirmed moderate-severe plaque psoriasis for at least 6 months before randomization.
* PASI scores≥12, IGA (mod 2011) scores ≥3 and BSA≥10% at screening and randomization.
* With indications for phototherapy or systemic therapy.
* Voluntarily sign informed consent.

Exclusion Criteria:

* Presented with pustular psoriasis, erythrodermic psoriasis，guttate psoriasis or psoriasis triggered by medicine at screening.
* Active persistent cutaneous inflammatory disease other than psoriasis at randomization.
* Treatment with phototherapy, including but not limited to ultraviolet A phototherapy (with or without psoralen), ultraviolet B phototherapy, or excimer laser within 4 weeks prior to randomization. Patients who are unwilling to avoid excessive UV exposure within 4 weeks prior to randomization and during this trial.
* Use of systemic treatment with anti-psoriasis non-biologic agents within 4 weeks prior to randomization, including but not limited to glucocorticoids, retinoids, cyclosporine, methotrexate, azathioprine, leflunomide, mycophenolate mofetil, tofacitinib, apremilast, traditional Chinese medicine/proprietary Chinese medicine, etc.
* Intra-articular glucocorticoid injection within 4 weeks or 5 drug half-lives (whichever is longer) prior to randomization.
* Topical anti-psoriasis treatment within 2 weeks prior to randomization.
* Prior treatment with the following biologic agents for the treatment of psoriasis within the specified time period prior to randomization: ustekinumab<6 months, Adalimumab, Etanercept, Infliximab, Golimumab, Guselkumab<12 weeks, Rituximab<12 months, or any other biological agent< 5 half lives.
* Prior treatment with anti-IL-17 antibody or anti-IL-17 receptor antibody.
* Meets any of the following at screening: haemoglobin<80 g/L, white blood cell<3×10E9/L, Neutrophils<1.5×10E9/L, platelet<75×10E9/L, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) and/or total bilirubin (TBiL)>2 times the upper limit of normal (ULN), serum creatinine (Scr)>1.5 ULN.
* History of inflammatory bowel disease or other disease with a high risk of perforation or other active autoimmune disease.
* Systemic infection or serious infection requiring hospitalization and/or intravenous anti-infective therapy within 4 weeks prior to randomization; any active infection within 2 weeks prior to randomization, with the exception of general upper respiratory tract infection.
* Have Received a live vaccine within 12 weeks prior to randomization, or plan to receive a live vaccine during the study or within 6 months after the last dose.
* Previously diagnosed or ongoing lymphoproliferative disorders. Malignant tumors within 5 years prior to screening, excluding squamous cell carcinoma of the skin or basal cell carcinoma or unflavored cervical cancer that have been cured after treatment.
* History of depression and/or any finding of suicidal ideation before randomization.
* Concomitant progressive or uncontrolled cardiovascular and cerebrovascular diseases, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, and neurological diseases, which are judged by the investigators to be inappropriate for participation in this study;
* Positive for any of the followings: hepatitis B virus surface antigen, hepatitis C virus antibody ,human immunodeficiency virus antibody, treponema pallidum antibody.
* Latent or active tuberculosis.
* Allergy to anti-IL-17 antibody active ingredients, excipients or latex.
* Pregnant or nursing women. Male or female patients who are unwilling to use effective contraception during the trial and for 5 months after the last dose
* Participated in other drug clinical trials within 3 months or 5 drug half-lives (whichever is longer) before screening.
* Any major surgery within 8 weeks prior to randomization, or planned major surgery during the study.
* History of recurrent drug abuse or unprescribed medication, or history of alcohol abuse.
* Other conditions judged by the investigator to be inappropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with PASI 75 at week 12. | week 12
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 75 is defined as at least a 75% reduction in PASI scores compared with the Baseline PASI scores.

SECONDARY OUTCOMES:
Proportion of patients with IGA (mod 2011) 0/1 at week 12. | week 12
  The modified version of Investigator's Global Assessment (IGA) wich was developed in 2011 (mod 2011) is a simple instrument providing a subjective evaluation of the overall severity of psoriasis. Erythema, induration, and scaling of psoriatic lesions are scored on a 5-point scale ranging from 0 (none) to 4 (severe) as the following:
  0=Clear (e.g., no signs of psoriasis, some post-inflammatory hyperpigmentation may be present) ; 1=Almost clear (e.g., no thickening, normal or pink coloration) ; 2=Mild (e.g., mild thickening, pink to light red coloration) ;3= Moderate (e.g., moderate thickening, dull to bright red) ; 4=Severe (e.g., severe thickening, bright to deep red) .
Proportion of patients with IGA (mod 2011) 0/1 at week 52. | week 52
  The modified version of Investigator's Global Assessment (IGA) wich was developed in 2011 (mod 2011) is a simple instrument providing a subjective evaluation of the overall severity of psoriasis. Erythema, induration, and scaling of psoriatic lesions are scored on a 5-point scale ranging from 0 (none) to 4 (severe) as the following:
  0=Clear (e.g., no signs of psoriasis, some post-inflammatory hyperpigmentation may be present) ; 1=Almost clear (e.g., no thickening, normal or pink coloration) ; 2=Mild (e.g., mild thickening, pink to light red coloration) ;3= Moderate (e.g., moderate thickening, dull to bright red) ; 4=Severe (e.g., severe thickening, bright to deep red) .
Proportion of patients with IGA (mod 2011) 0 at week 12. | week 12
  The modified version of Investigator's Global Assessment (IGA) wich was developed in 2011 (mod 2011) is a simple instrument providing a subjective evaluation of the overall severity of psoriasis. Erythema, induration, and scaling of psoriatic lesions are scored on a 5-point scale ranging from 0 (none) to 4 (severe) as the following:
  0=Clear (e.g., no signs of psoriasis, some post-inflammatory hyperpigmentation may be present) ; 1=Almost clear (e.g., no thickening, normal or pink coloration) ; 2=Mild (e.g., mild thickening, pink to light red coloration) ;3= Moderate (e.g., moderate thickening, dull to bright red) ; 4=Severe (e.g., severe thickening, bright to deep red) .
Proportion of patients with IGA (mod 2011) 0 at week 52. | week 52
  The modified version of Investigator's Global Assessment (IGA) wich was developed in 2011 (mod 2011) is a simple instrument providing a subjective evaluation of the overall severity of psoriasis. Erythema, induration, and scaling of psoriatic lesions are scored on a 5-point scale ranging from 0 (none) to 4 (severe) as the following:
  0=Clear (e.g., no signs of psoriasis, some post-inflammatory hyperpigmentation may be present) ; 1=Almost clear (e.g., no thickening, normal or pink coloration) ; 2=Mild (e.g., mild thickening, pink to light red coloration) ;3= Moderate (e.g., moderate thickening, dull to bright red) ; 4=Severe (e.g., severe thickening, bright to deep red) .
Proportion of patients with PASI 50 at week 12. | week 12
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 50 is defined as at least a 50% reduction in PASI scores compared with the Baseline PASI scores.
Proportion of patients with PASI 75 at week 52. | week 52
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 75 is defined as at least a 75% reduction in PASI scores compared with the Baseline PASI scores.
Proportion of patients with PASI 90 at week 12. | week 12
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 90 is defined as at least a 90% reduction in PASI scores compared with the Baseline PASI scores.
Proportion of patients with PASI 90 at week 52. | week 52
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 90 is defined as at least a 90% reduction in PASI scores compared with the Baseline PASI scores.
Proportion of patients with PASI 100 at week 12. | week 12
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 100 is defined as complete remission.
Proportion of patients with PASI 100 at week 52. | week 52
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 100 is defined as complete remission..
Change from baseline in DLQI at week 52 | week 52.
  The Dermatology Life Quality Index (DLQI) is the most commonly used dermatology-specific quality of life (QOL) measure in clinical trials of skin diseases. It consists of 10 questions concerning dermatologic patients' perception of the impact of skin diseases on different aspects of their QOL over the last week. The items of the DLQI encompass aspects such as symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale: 0=not at all/not relevant , 1=a little, 2=a lot, and 3=very much. Scores of individual items are added to yield a total score (0-30). A DLQI score of 0 and 1 means no impact ona patient's QOL whereas a score of 2~5, 6~10, 11~20, and 21~30 indicates a small, moderate, large, and an extremely large effect on patient's QOL, respectively.
Change from baseline in PASI at week 52 | week 52.
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.
Change from baseline in IGA (mod 2011) at week 52 | week 52.
  The modified version of Investigator's Global Assessment (IGA) wich was developed in 2011 (mod 2011) is a simple instrument providing a subjective evaluation of the overall severity of psoriasis. Erythema, induration, and scaling of psoriatic lesions are scored on a 5-point scale ranging from 0 (none) to 4 (severe) as the following:
  0=Clear (e.g., no signs of psoriasis, some post-inflammatory hyperpigmentation may be present) ; 1=Almost clear (e.g., no thickening, normal or pink coloration) ; 2=Mild (e.g., mild thickening, pink to light red coloration) ;3= Moderate (e.g., moderate thickening, dull to bright red) ; 4=Severe (e.g., severe thickening, bright to deep red) .
Change from baseline in BSA at week 52 | week 52
  Body Surface Area (BSA) score is an important indicator for calculating the overall skin lesion area of psoriasis. BSA ≈1% refers to the area of the skin lesion as the size of a palm, and the estimation of the skin lesion area in this method can roughly assess the severity of the disease.
Incidence of adverse events | week 52
  Number of patients reporting at least one adverse event in the study. An adverse event is defined as any untoward medical occurrence in a clinical trial participant graded according to the common terminology criteria for adverse events (CTCAE) v.5.0 criteria,including clinically-significant changes in physical examinations, laboratory safety tests, ECG and vital signs
Immunogenicity | week 52
  Percentage of anti-drug antibody and neutralizing antibody in the study. Subjects with a positive antibody response to CMAB015 or Secukinumab were determined to test neutralizing antibody.

OTHER OUTCOMES:
AUC0-t | week 52
  AUC0-t, the area under the concentration-time curve from time zero to the time of the last quantifiable concentration, will be analyzed using a non-atrioventricular model.
AUC0-inf | week 52
  AUC0-inf, the area under the concentration-time curve from time zero to infinity, will be analyzed using a non-atrioventricular model.
Half time | week 52
  Half time will be analyzed using a non-atrioventricular model.
Cmax | week 52
  Cmax is the maximum concentration.
Tmax | week 52
  Tmax is the time of the maximum concentration.
Clearance Rate | week 52
  Clearance rate will be analyzed using a non-atrioventricular model.
Apparent Volume of Distribution | week 52
  Apparent Volume of Distribution will be analyzed using a non-atrioventricular model.

CONTACTS AND LOCATIONS:
Overall Officials: Jin h Xu, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China